CLINICAL TRIAL: NCT03902379
Title: Web-Based Coping and Communication Skills Intervention for Women Who Are Newly Diagnosed With Gynecological Cancer: A Pilot Study
Brief Title: Web-Based Coping and Communication Skills Intervention in Improving Psychological Adaptation in Patients With Gynecological Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was never initiated, no patients were enrolled. It has been closed with the IRB.
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Sharon Manne, PhD, Professor of Medicine, Rutgers Cancer Institute of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro20160000637; NCI-2017-02300 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); Pro20160000637; 131602 (Other: Rutgers Cancer Institute of New Jersey); P30CA072720 (NIH)
Record Dates: First submitted 2018-07-06; First posted 2019-04-04 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Endometrial Carcinoma; Stage 0 Fallopian Tube Cancer AJCC v7; Stage I Fallopian Tube Cancer AJCC v6 and v7; Stage I Ovarian Cancer AJCC v6 and v7; Stage IA Fallopian Tube Cancer AJCC v6 and v7; Stage IA Ovarian Cancer AJCC v6 and v7; Stage IB Fallopian Tube Cancer AJCC v6 and v7; Stage IB Ovarian Cancer AJCC v6 and v7; Stage IC Fallopian Tube Cancer AJCC v6 and v7; Stage IC Ovarian Cancer AJCC v6 and v7; Stage II Cervical Cancer AJCC v7; Stage II Fallopian Tube Cancer AJCC v6 and v7; Stage II Ovarian Cancer AJCC v6 and v7; Stage II Uterine Corpus Cancer AJCC v7; Stage IIA Cervical Cancer AJCC v7; Stage IIA Fallopian Tube Cancer AJCC v6 and v7; Stage IIA Ovarian Cancer AJCC V6 and v7; Stage IIA1 Cervical Cancer AJCC v7; Stage IIA2 Cervical Cancer AJCC v7; Stage IIB Cervical Cancer AJCC v6 and v7; Stage IIB Fallopian Tube Cancer AJCC v6 and v7; Stage IIB Ovarian Cancer AJCC v6 and v7; Stage IIC Fallopian Tube Cancer AJCC v6 and v7; Stage IIC Ovarian Cancer AJCC v6 and v7; Stage III Cervical Cancer AJCC v6 and v7; Stage III Fallopian Tube Cancer AJCC v7; Stage III Ovarian Cancer AJCC v6 and v7; Stage III Primary Peritoneal Cancer AJCC v7; Stage III Uterine Corpus Cancer AJCC v7; Stage IIIA Cervical Cancer AJCC v6 and v7; Stage IIIA Fallopian Tube Cancer AJCC v7; Stage IIIA Ovarian Cancer AJCC v6 and v7; Stage IIIA Primary Peritoneal Cancer AJCC v7; Stage IIIA Uterine Corpus Cancer AJCC v7; Stage IIIB Cervical Cancer AJCC v6 and v7; Stage IIIB Fallopian Tube Cancer AJCC v7; Stage IIIB Ovarian Cancer AJCC v6 and v7; Stage IIIB Primary Peritoneal Cancer AJCC v7; Stage IIIB Uterine Corpus Cancer AJCC v7; Stage IIIC Fallopian Tube Cancer AJCC v7; Stage IIIC Ovarian Cancer AJCC v6 and v7; Stage IIIC Primary Peritoneal Cancer AJCC v7; Stage IIIC Uterine Corpus Cancer AJCC v7; Stage IIIC1 Uterine Corpus Cancer AJCC v7; Stage IIIC2 Uterine Corpus Cancer AJCC v7; Stage IV Cervical Cancer AJCC v6 and v7; Stage IV Fallopian Tube Cancer AJCC v6 and v7; Stage IV Ovarian Cancer AJCC v6 and v7; Stage IV Primary Peritoneal Cancer AJCC v7; Stage IV Uterine Corpus Cancer AJCC v7; Stage IVA Cervical Cancer AJCC v6 and v7; Stage IVA Uterine Corpus Cancer AJCC v7; Stage IVB Cervical Cancer AJCC v6 and v7; Stage IVB Uterine Corpus Cancer AJCC v7; Uterine Carcinosarcoma; Uterine Corpus Sarcoma
MeSH Terms: conditions — Endometrial Neoplasms; Fallopian Tube Neoplasms; Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive Care (CCI intervention) (Experimental): Patients complete 3 modules of online CCI intervention.
  Interventions: Other: Internet-Based Intervention; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Other: Survey Administration

INTERVENTIONS:
Other: Internet-Based Intervention — Receive CCI intervention
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Other: Survey Administration — Ancillary studies

SUMMARY:
This pilot clinical trial studies how well web-based coping and communication skills intervention works in improving psychological adaptation in patients with gynecological cancer. Web-based intervention, such as coping and communication skills intervention, may help doctors to get a better understanding of ways to help gynecological cancer patients cope with their cancer experience.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To examine the feasibility and acceptability of an online coping and communication skills intervention (CCI).

II. To collect pilot data on the impact of online CCI on global and cancer-specific distress.

OUTLINE:

Patients complete 3 modules of online CCI intervention.

After completion of study, patients are followed up at 2 months.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed with any stage of primary ovarian cancer, primary peritoneal cancer, or primary fallopian tube cancer in the past 6 months
* Newly diagnosed with high grade stage 2, any grade stage 3 or higher endometrial cancer in the past 6 months
* Newly diagnosed with stage 2 or higher cervical cancer within the past 6 months
* Newly diagnosed with any stage uterine cancer (both sarcoma and carcinosarcoma) in the past 6 months
* At the time of recruitment the patient is on active treatment defined as either currently receiving chemotherapy or radiation or less than 6 months post-cancer surgery
* At the time of recruitment, a Karnofsky performance status of 80 or above or an Eastern Cooperative Oncology Group (ECOG) (80) score of 0 or 1
* English speaking
* Has internet access
* Must give informed consent within 6 months of diagnosis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-07-27 (Actual); Primary Completion 2020-05-31 (Estimated); Study Completion 2020-05-31 (Estimated)

PRIMARY OUTCOMES:
Examine feasibility of an online CCI as defined by participant's evaluation of the online intervention | Up to 2 months
  Will define feasibility/acceptability as participant's evaluation of the online intervention using both qualitative and quantitative methods. Will summarize participant?s feedback by their overall impressions, the ease of use, how much the web intervention kept their attention, how much they liked the program, feedback about how the program looked, suggestions on how to improve the look, their satisfaction with the program and why, how useful they found the program and why, how easy the information was to understand and why, to what degree they think it would make them more confident in coping with cancer, what the most and least helpful components of the program were, what aspects if any were confusing, evaluation of places where navigation were unclear, and anything they would like to add to the program.

SECONDARY OUTCOMES:
Changes in psychological adaptation- Beck Depression Inventory (BDI) | Baseline up to 2 months
  Pre-post changes in the(BDI) scales will be examined. BDI has 21 items and scores range 0-63
Changes in psychological adaptation-Mental Health Inventory (MHI) | Baseline up to 2 months
  Pre-post changes in the (MHI) scales will be examined t-tests. 38-item MHI measure used
Changes in psychological coping | Baseline up to 2 months
  Pre-post changes in the Impact of Event Scale (IES) scales will be examined using t-tests.
Examine acceptability of an online CCI | Up to 2 months
  Will define acceptability as participant's evaluation of the online intervention using both qualitative and quantitative methods. Will summarize participant?s feedback by their overall impressions, the ease of use, how much the web intervention kept their attention, how much they liked the program, feedback about how the program looked, suggestions on how to improve the look, their satisfaction with the program and why, how useful they found the program and why, how easy the information was to understand and why, to what degree they think it would make them more confident in coping with cancer, what the most and least helpful components of the program were, what aspects if any were confusing, evaluation of places where navigation were unclear, and anything they would like to add to the program.

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Manne, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (1):
- Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey, United States